CLINICAL TRIAL: NCT02292199
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Sympathetic and Parasympathetic Nervous System in Patients With Hypertension: a Randomized Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation on Nervous System in Patients With Hypertension.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Effects of transcutaneous electrical nerve stimulation on sympathetic and parasympathetic nervous system in patients with hypertension: a randomized clinical trial, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYPERTENSIONTENS
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Cardiovascular Diseases
Keywords: Hypertension; TENS; Sympathetic and Parasympathetic nervous system
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TENS High Frequency 100 Hz (Experimental): TENS was applied for thirty minutes, with the frequency defined according to randomization. The intensity of the current was delivered at sensory-level intensity, adjusted every 5 minutes by the sensory threshold, during the 30 minutes as tolerated by each subject, but without motor contraction or pain reported by the subject.
  Interventions: Device: TENS High Frequency
- TENS Low Frequency 4 Hz (Active Comparator): TENS was applied for thirty minutes, with the frequency defined according to randomization. The intensity of the current was delivered at sensory-level intensity, adjusted every 5 minutes by the sensory threshold, during the 30 minutes as tolerated by each subject, but without motor contraction or pain reported by the subject.
  Interventions: Device: TENS Low Frequency
- TENS Placebo (Placebo Comparator): The placebo group received an active current for 30 seconds, and then gradually decreased for 15 seconds to not pass any current. This approach aims at masking the investigator and subject (RAKEL et al., 2010).
  Interventions: Device: TENS Placebo

INTERVENTIONS:
Device: TENS High Frequency — TENS high frequency (100 Hz / 200μs) was applied in bilateral paravertebral region of the T1 segment of the thoracic spine at L2 lumbar spine. The intensity of the current was delivered at sensory-level intensity, adjusted every 5 minutes by the sensory threshold, during the 30 minutes as tolerated by each subject, but without motor contraction or pain reported by the subject.
  Arms: TENS High Frequency 100 Hz
Device: TENS Low Frequency — TENS low frequency (4 Hz / 200μs) was applied in bilateral paravertebral region of the T1 segment of the thoracic spine at L2 lumbar spine. The intensity of the current was delivered at sensory-level intensity, adjusted every 5 minutes by the sensory threshold, during the 30 minutes as tolerated by each subject, but without motor contraction or pain reported by the subject.
  Arms: TENS Low Frequency 4 Hz
Device: TENS Placebo — TENS was applied in bilateral paravertebral region of the T1 segment of the thoracic spine at L2 lumbar spine. The placebo group received an active current for 30 seconds, and then gradually decreased for 15 seconds to not pass any current. This approach aims at masking the investigator and subject (RAKEL et al., 2010).
  Arms: TENS Placebo

SUMMARY:
Hypertension has high prevalence and poor control rates and is considered one of the major modifiable risk factors for cardiovascular system diseases, and one of the most important public health problems. The imbalance of the autonomic cardiovascular control, which can be considered as a major etiologic factor in the development of essential hypertension is characterized by increased sympathetic activity and reduced parasympathetic activity possible.

Cardiovascular disease is the leading cause of death and disability in the world and autonomic imbalance is associated with several pathological conditions, and may be a final common pathway for the increased morbidity and mortality of cardiovascular diseases. In this sense, the heart rate variability (HRV) is a quantitative marker of sympathetic and parasympathetic activity, which can be used to assess disease and mortality as a noninvasive technique.

TENS is a noninvasive therapeutic modality, easy to handle, it has no side effects or interactions with medications being used for the relief of pain by sensory stimulation through peripheral nerves and mainly for control and treatment of acute and chronic pain . Research on the effect of TENS on the sympathetic and parasympathetic nervous system activity remain controversial, especially regarding the parameters to use.

The aim of this study is to investigate the effects of TENS on the sympathetic and parasympathetic nervous system in patients with hypertension by heart rate variability and blood pressure variability.

This is a randomized clinical trial, double blind, where hypertensive patients were randomized to three groups: high-frequency TENS (100 Hz) n = 20, low frequency TENS (4 Hz) n = 20 and n = 20 placebo. Evaluations will be made in a single session. The results will be assessed by a blinded investigator and randomization will be done electronically.

It is expected to evaluate how often TENS exerts more influence in the modulation of sympathetic and parasympathetic system.

DETAILED DESCRIPTION:
Data collection was performed at the Laboratory of Clinical Investigation (LIC) Institute of Cardiology. Initially, patients rested for 30 minutes, and during this period has been completed the evaluation form with the identification data and questions about the patient's clinical status, such as checking blood pressure, weight and height.

Patients were randomized to group of high frequency (100 Hz / 200μs), low frequency (4 Hz / 200μs) or placebo. The placebo group received an active current for 30 seconds, and then gradually decreased for 15 seconds to not pass any current. This approach aims at masking the investigator and subject (RAKEL et al., 2010). Eligible subjects were randomly assigned in blocks, by electronic randomization (www.randomization.com).

The adhesive electrodes were used, size 9x5 cm, placed in bilateral paravertebral region of the T1 segment of the thoracic spine at L2 lumbar spine. Before the application of TENS (IBRAMED®), the skin was cleaned in place of the current application with alcohol to avoid any barrier conduction of electrical current.

The sessions took place at the same time of the day, throughout the protocol, the participants were comfortably accommodated in an acclimatized room (23ºC) in a supine position, head elevation of 30º with knees resting on a wedge. All the participants were forbidden to perform exhaustive exercises and intake caffeine at least two hours before the intervention and instructed to have a meal before the assessment.

TENS was applied for thirty minutes, with the frequency defined according to randomization. The intensity of the current was delivered at sensory-level intensity, adjusted every 5 minutes by the sensory threshold, during the 30 minutes as tolerated by each subject, but without motor contraction or pain reported by the subject.

The analysis of autonomic control was performed by means of a sensor placed on the middle finger, and connected to the Finapres (Ohmeda 2300, Colorado, USA) by recording beat to beat. Then, the conversion signal was performed using the powerlab (LAB chart). The analysis will be performed using the software Kubios.

ELIGIBILITY:
Inclusion Criteria:

Previous Hypertension diagnosis, systolic blood pressure (SBP) > 140 mm Hg and/or diastolic blood pressure (DBP) >90 mm Hg and clinical stability with no change in medications for at least 2 months preceding the study.

Exclusion Criteria:

Presence of any comorbidity such as diabetes; congestive heart failure; unstable angina; myocardial infarction; acute inflammation; peripheral vascular disease; associated neurological disease; acute respiratory illness; infectious disease or fever; cardiac pacemaker; unstable ventricular arrhythmia; active smokers; obesity; musculoskeletal disease in the lower limbs; changes in the electrocardiogram; smoker; treatment with beta blockers, steroids, hormones or chemotherapy or change in drug therapy were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 2 Hours
  For the analysis of heart rate variability (HRV), the time of RR intervals obtained from continuous ECG signal recorded by Finapres device (Ohmeda 2300, Colorado, USA) series. The time series of RR will be analyzed in the time and frequency and variability parameters and autonomic balance will be obtained. In the time domain we calculate the mean values of RR intervals, standard deviation and the square root of the sum of the square of successive differences (rMSSD). The acquisition of electrocardiogram signal (ECG) was performed immediately before and after the interventions for a 10-minute period, with the subject at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, Phd, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Rodrigo Della Méa Plentz, Porto Alegre, Rio Grande do Sul, Brazil